CLINICAL TRIAL: NCT01409148
Title: Radioimmunoimaging (PET/CT) of Patients With AL Amyloidosis Using the 124I-Labeled Amyloid-Reactive Monoclonal Antibody Mu 11-1F4
Brief Title: Radioimmunoimaging of AL Amyloidosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alan Solomon, Professor of Medicine, University of Tennessee
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2625A; FD-R-003420-01-A1
Record Dates: First submitted 2011-07-28; First posted 2011-08-04 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2011-08

CONDITIONS: AL Amyloidosis
Keywords: Radioimmunoimaging; AL Amyloidosis; PET/CT
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I-124 Mu 11-1F4 sterile injection (Other): Single arm study
  Interventions: Biological: 124I-labeled monoclonal antibody Mu 11-1F4

INTERVENTIONS:
Biological: 124I-labeled monoclonal antibody Mu 11-1F4 — Single infusion of radiolabeled antibody: 2mCi (1 mg)

SUMMARY:
The purpose of the study is to determine the capability of a radiolabeled amyloid-reactive monoclonal antibody to document the presence and distribution of amyloid deposits by PET/CT imaging in patients with AL amyloidosis.

DETAILED DESCRIPTION:
To be eligible for this study, patients must have a confirmed diagnosis of AL amyloidosis without significant cardiac (New York Heart Association class IV) disease and not be on kidney dialysis. Additionally, after testing, their blood must not contain antibodies to mouse proteins. The study requires an intravenous infusion, over 10 minutes, of the radiolabeled antibody, followed 48 hours later by a PET/CT scan. A repeat scan is done 5 or 7 days after infusion of the antibody. A 5 ml blood specimen needs to be furnished 4 and 8 weeks after the antibody infusion.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of AL Amyloidosis

Exclusion Criteria:

* New York Heart Association class IV
* patient on renal dialysis
* serum antibodies to mouse protein

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Radioimmunoimaging of AL amyloid deposits | 36 months

SECONDARY OUTCOMES:
Imaging of amyloid deposits as determined by PET/CT | 10-14 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States

REFERENCES:
- See also: Amyloid research foundation — http://www.ARFAmyloid@aol.com